CLINICAL TRIAL: NCT01396967
Title: The Efficiency of a New Device for Performing Capsulorhexis in Cataract Surgery
Brief Title: Trying a New Device for Performing Capsulorhexis in Cataract Surgery Surgery
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Joseph Pikkel MD, Ziv Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ZIV-0065-10
Record Dates: First submitted 2011-07-13; First posted 2011-07-19 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Eye Disease; Cataract
Keywords: capsulorhexis
MeSH Terms: conditions — Eye Diseases; Cataract | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: surgery — cataract surgery
  Other Names: V.R.hexis-1

SUMMARY:
During cataract operations a capsulorhexis is being performed. This is done in order to enable the removal of lens material while keeping the capsule intact in order to put inside the lens capsule an artificial intra ocular lens.

The capsulorhexis must be round and with regular edge and no tears. While performing a cataract surgery we use phako emulsification machine that sends an ultrasonic wave that creaks the lens nucleus and at the same time irrigates the anterior chamber of the eye and sucks the fluid and the lens material of the creaked lens.

The round shape and the regularity of the capsulorhexis are a must in these surgeries since the lens capsule must stay intact and stable in order to enable the phacoemulsification and the implant of the artificial lens.

Today capsulorhexis are done with a bent needle or with special forceps; the act of capsulorhexis is delicate, sometime un predicted and difficult to teach. The learning curve is relatively long and difficult.

The proposed device enables a capsulorhexis which is round and has regular edges, done almost automatically and is predicted. The learning curve is short and easy. The capsulorhexis is done through the original operating wound with no need to widen it.

DETAILED DESCRIPTION:
Planed Procedure

20 patients will be tested in this trail.

Consecutive patients that have senile cataract will be examined preoperatively as is done usually and the data of the examination will be collected/ a special attention will be given to the type of cataract and lens stability.

Systemic diseases will not be considered as exclusion criteria.

Patients with dens or mature cataract will be excluded.

Patients will be explained about the new device and those who will agree will sign a consent form.

During the cataract surgery all steps will be done as usually except of the capsulorhexis which will be done by using the new device.

The capsulorhexis will be photographed for further evaluation by a microscope camera.

After the operation the surgeon will record his impression about the convenience of using the new device, the shape and form of the capsulorhexis and its stability and any other relevant information.

Post operative follow up will be done as usually, one day, one week, 3 weeks and six weeks after operation. The results of those examinations will be recorded and collected with special attention of IOL stability, the shape of capsulorhexis and intra ocular post operative inflammation if will occur.

The data, including the surgeons' comments, shape and form of capsulorhexis IOL stability and the rest will be collected and processed.

In case in which the use of the device will not perform a round and regular capsulorhexis, or instability of the capsule will occur or a un predicted intraocular inflammation will be seen the trail will be stopped immediately

ELIGIBILITY:
Inclusion Criteria:

* senile cataract

Exclusion Criteria:

* dens or mature cataract trauma congenital instability of the lens(phacodonesis,TXF)

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
capsulorhexis must be round and with regular edge and no tears | Post operative follow up will be done as usually, one day, one week, 3 weeks and six weeks after operation
  As the title of this experiment:"The trying a new device for performing capsulorhexis in cataract surgery".Becuase we are not changing the protocol of Cataract surgery,the outcome measure of this experiment is the efficiency of this device, the safety and the simplicity of the use the device inorder to give a simple and safe solution for capsulorhexis.Therefor the outcome measure will be IOL stability, the shape of capsulorexis and intra ocular post operative inflammation if will occur. The trail is not comparative.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Pikkel, Md, Principal Investigator — Ziv Medical Center Sefat Israel
Locations (1):
- Ziv Medical Center, Safed, Israel